CLINICAL TRIAL: NCT04900766
Title: A Multicenter, Open-label, Phase Ib Study of Mitoxantrone Hydrochloride Liposome Injection in Subjects With Advanced Bone and Soft Tissue Sarcoma Who Has Failed At Least One Prior Line of Therapy
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection in Subjects With Advanced Bone and Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor has adjusted its R&D strategy.
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-019
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Unresectable or Metastatic Bone and Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): Subjects with unresectable or metastatic bone and soft tissue sarcoma will receive 20 mg/m2 Mitoxantrone Hydrochloride Liposome injection every 21 days (a cycle) for a maximum of 6 cycles.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome Injection — 20 mg/m2, IV, on day 1 of each 21-day cycle (q3w).

SUMMARY:
This is a multicenter, open-label, phase Ib study to evaluate the safety and efficacy of Mitoxantrone Hydrochloride Liposome in subjects with unresectable or metastatic bone and soft tissue sarcoma who has failed at least one prior line of therapy.

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase Ib study to evaluate the safety and efficacy of Mitoxantrone Hydrochloride Liposome in subjects with unresectable or metastatic bone and soft tissue sarcoma who has failed at least one prior line of therapy. About 50 subjects will be recruited in this study. The subjects will receive Mitoxantrone Hydrochloride Liposome 20 mg/m2 by an intravenous infusion (IV), every 21 days (q3w, 1 cycle). All the subjects will receive the treatment until disease progression, intolerable toxicity, death, or withdrawal by investigator or subject decision (a maximum of 6 cycles).

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects fully understand and voluntarily participate in this study and sign informed consent; 2. Age ≥18 years, without gender limitation; 3. Histologically confirmed diagnosis of bone or soft tissue sarcoma; 4. Metastatic or unresectable bone or soft tissue sarcoma that has failed at least one prior line of therapy; 5. At least one measurable lesion according to RECIST v1.1; 6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; 7. Adequate organ function defined as:

  * Absolute neutrophil count (ANC) ≥1.5 x109/L (No G-CSF treatment within 1 week prior to the laboratory test);
  * Hemoglobin ≥ 110 g/L (No red blood cell transfusion within 1 week prior to the laboratory test);
  * Platelet count ≥ 100 x 109/L (No platelet transfusion within 1 week prior to the laboratory test);
  * Creatinine ≤1.5 x upper limit of normal (ULN);
  * Total bilirubin ≤1.5 x ULN (≤3.0 x ULN for liver metastasis);
  * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 3 x ULN (≤5.0 x ULN for liver metastasis);
  * Coagulation: Prothrombin time (PT) or International Normalization Ratio (INR) ≤1.5 x ULN (≤3.0 x for those receiving anticoagulant drugs such as warfarin); 8. Female subjects must have a urine or blood HCG negative test (except for menopause and hysterectomy); 9. Subjects and their partners must agree to use effective contraceptive measures during the study until 6 months after the end of the last dose.

Exclusion Criteria:

* 1. History of severe allergy to mitoxantrone hydrochloride or liposomal drugs; 2. Cerebral or meningeal metastases; 3. History of allogeneic organ transplantation or allogeneic bone marrow transplantation; 4. Life expectancy < 12 weeks; 5. Subjects with chronic hepatitis B (HBsAg or HBcAb positive with HBV DNA ≥ 1000 IU/mL), hepatitis C (HCV antibody positive with HCV RNA above the lower limit of detection of the study center), or human immunodeficiency virus (HIV) antibody positive;; 6. AEs from the previous treatment > Grade 1 based on CTCAE (except for the toxicity without safety risk judged by the investigator, such as alopecia, hyperpigmentation); 7. Active bacterial, fungal or viral infections that require systemic treatment within 1 week prior to the first dose; 8. Local or systemic anticancer treatment within 4 weeks prior to the first dose (within 2 weeks prior to dosing for traditional Chinese medicine or proprietary Chinese medicine); 9. Enrolled in any other clinical trials within 4 weeks prior to the first dose; 10. Thrombosis or thromboembolism within 6 months prior to screening; 11. History of, or known additional malignant tumor within 3 years, except for locally curable tumors that have been cured, such as basal or squamous cell skin cancer or in situ prostate, cervical or breast cancer; 12. Impaired cardiac function or serious cardiac disease:

  * Long QTc syndrome or QTc interval > 480 ms;
  * Complete left bundle branch block, II-III degree atrioventricular block;
  * Severe, uncontrolled arrhythmias requiring pharmacological treatment;
  * History of chronic congestive heart failure, NYHA ≥ grade 3;
  * Cardiac ejection fraction < 50% within 6 months prior to screening;
  * Heart valve disease with CTCAE ≥ grade 3;
  * Uncontrollable hypertension (defined as a measured systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg under pharmacological control);
  * ECG evidence of myocardial infarction, unstable angina, history of severe pericardial disease, and acute ischemic or severe conduction system abnormalities within 6 months prior to screening; 13. Previous treatment with adriamycin or other anthracyclines, and the total cumulative dose of prior adriamycin or equivalent is >350 mg/m2.

    14. Pregnant or lactating female; 15. Serious and/or uncontrolled medical condition that, in the judgment of the investigator, may affect the patient's participation in this study (including, but not limited to: diabetes not effectively controlled, kidney disease requiring dialysis, severe liver disease, life-threatening autoimmune and bleeding disorders, substance abuse, neurological disorders, etc.); 16. Not suitable for this study as decided by the investigator due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
TEAEs | From the initiation of the first dose to 28 days after the last dose
  Treatment-emergent adverse events

SECONDARY OUTCOMES:
ORR | up to 36 months
  Overall response rate
DoR | up to 36 months
  Duration of response
DCR | up to 36 months
  disease control rate
PFS | up to 36 months
  progression-free survival
OS | up to 36 months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Niu, Bachelor, Principal Investigator — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No